CLINICAL TRIAL: NCT00059358
Title: Pharmacological Interactions Between Zidovudine and Ribavirin in HCV-HIV Co-Infected Patients Treated With Rebetron or Peg-Intron Plus Ribavirin
Brief Title: Zidovudine Levels in HIV Infected Patients Being Treated for HCV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jose F. Rodriguez, PhD, MSC-UPR
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI09141-01A1; 5R01AI049141-02 (NIH)
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV; HCV; Ribavirin; Interferon; Co-infection; Treatment experienced
MeSH Terms: conditions — HIV Infections; Hepatitis C; Coinfection | interventions — Ribavirin; Interferon alpha-2; peginterferon alfa-2b

ARMS (1):
- 1 (Experimental): Participants will begin receive either Rebetron or PEG-Intron plus ribavirin therapy from Weeks 2 through 48
  Interventions: Drug: Ribavirin plus interferon alfa-2b; Drug: Ribavirin; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: Ribavirin plus interferon alfa-2b — Oral tablets taken daily
Drug: Ribavirin — Oral tablet taken daily
Drug: Peginterferon alfa-2b — Subcutaneous injection

SUMMARY:
This study will test the amount of anti-HIV drugs in the blood cells of HIV-infected patients who are also being treated for hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
An estimated 50,000 people in Puerto Rico are infected with HCV. HIV and HCV have similar routes of transmission, and HCV co-infection occurs in 8% to 23% of HIV infected patients. Researchers have shown that treatment for HCV with Rebetron (ribavirin plus interferon alfa-2b) significantly decreases HCV viral load without affecting HIV viral load. However, measurements of intracellular levels of the active forms of zidovudine (ZDV-MP and ZDV-TP) were not performed. Such measurements are needed to provide a more rational basis for dosing in HIV/HCV co-infected patients. This study will investigate the intracellular exposure to active ZDV metabolites prior to and after treatment with Rebetron or treatment with PEG-Intron (pegylated interferon) and ribavirin.

Participants in this study will remain on their usual antiretroviral regimen; no changes may be made to that regimen for the first 4 weeks of the study. Upon study entry, participants will have intracellular pharmacokinetic studies. During Week 2, participants will start either Rebetron or PEG-Intron plus ribavirin therapy, will have intracellular pharmacokinetic studies, and will undergo liver biopsy. Additional intracellular pharmacokinetic studies will be performed at Weeks 12 and 24. Rebetron or PEG-Intron plus ribavirin will be given for 48 weeks. A second liver biopsy will be performed 24 weeks after discontinuing Rebetron or PEG-Intron plus ribavirin therapy. Participants will be followed for 72 weeks.

ELIGIBILITY:
Inclusion Criteria

* HCV-infected
* HIV-1 infection
* CD4 cell count > 200 cells/mm³ within 30 days prior to study entry
* HIV RNA < 400 copies/ml within 90 days of study entry
* Use of zidovudine, lamivudine, and any PI and/or NNRTI
* ANC value >= 1,500 ml³ within 30 days of study entry
* Weight > 50 kg (110 lbs) for women and > 60 kg (132 lbs) for men
* Acceptable methods of contraception
* Ability and willingness to complete the Baseline Adherence Questionnaire
* Documentation of adherence confirmed by the Baseline Adherence Questionnaire and certified by the study officials

Exclusion Criteria

* Previous ribavirin therapy
* More than 2 months of interferon therapy
* Current use of any NRTI other than ZDV and 3TC
* Hepatitis B surface antigen positive
* Infectious, autoimmune, tumoral, biliary, or vascular liver disease
* Alcohol consumption of more than 50 g/day
* Current use of intravenous drugs
* Hemoglobin levels < 10 gm/dl
* Methadone use
* Chemotherapy
* Certain medications
* Acute opportunistic or bacterial infection requiring therapy at the time of enrollment
* Hemoglobinopathy (e.g., thalassemia) or any other cause of tendency to hemolysis
* Psychiatric disorders, severe depression, history of suicide attempts, or suicidal ideation
* Renal disease requiring dialysis
* Significant coronary diseases or two or more risk factors for coronary diseases, such as > 55 years old, hypertension, and cholesterol > 250 mg/dl
* Any clinically significant diseases (other than HIV and HCV infection) that, in the opinion of study officials, would compromise the outcome of this study
* Pregnancy
* Participation in blinded clinical trial

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2001-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Steady state area under the concentration time curve (AUC) between 0 and 12 hours of zidovudine (ZDV)-MP, ZDV-TP, and dTTP in PBMCs from HIV and hepatitis C virus (HCV) coinfected patients before and after peginterferon alfa-2b with or without ribavirin | Throughout study
Systemic exposure (AUC over 0 to 12 hours) of nelfinavir before and after peginterferon alfa-2b with or without ribavirin in HIV and HCV coinfected patients | Throughout study
Effect of peginterferon alfa-2b with or without ribavirin in HCV RNA viral titers, alanine aminotransferase (ALT) levels, CD4+, and HIV-RNA viral titers in HIV and HCV coinfected patients | Through Week 48
Effect of peginterferon alfa-2b with or without ribavirin on liver histology | At Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Jose F. Rodriguez, PhD, Principal Investigator — MSC-UPR; Jorge L. Santana, MD, Principal Investigator — MSC-UPR
Locations (1):
- UPR Adult ACTU, San Juan, Puerto Rico